CLINICAL TRIAL: NCT05115591
Title: The Use of Ultrasound to Predict a Difficult Spinal Anesthesia: a Prospective Single-blind Observational Study
Brief Title: Ultrasound Predictors of Difficult Spinal Anesthesia
Acronym: SPINAL-US
Status: Completed | Type: Observational
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Giuseppe Pascarella, Principal Investigator, Campus Bio-Medico University
Other Study IDs: 19.21 OSS
Record Dates: First submitted 2021-10-30; First posted 2021-11-10 (Actual); Last update posted 2021-11-18 (Actual); Status verified 2021-11

CONDITIONS: Anesthesia; Procedural Complication
Keywords: Spinal Anesthesia; Ultrasound
MeSH Terms: interventions — Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Spinal Ultrasound — Spinal Ultrasound is performed by an observer who records ultrasound characteristics of the intervertebral space chosen by the anesthetist who will practice spinal anesthesia
Procedure: Spinal Anesthesia — Spinal anesthesia is performed by an anesthetist after the observer recorded ultrasound characteristics of the intervertebral space chosen by the anesthetist, who is blinded to the ultrasound evaluation.

SUMMARY:
This prospective observational study aims to investigate about the efficacy of spine ultrasound in predicting difficult spinal anesthesia

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing spinal anesthesia for elective surgery
* ASA physical status score < 4

Exclusion Criteria:

* Contraindications to regional anesthesia
* ASA physical status score ≥ 4
* Patient's refusal or inability to sing the informed consent
* Previous spine surgery affecting the intervertebral space chosen for spinal anesthesia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing spinal anesthesia for elective orthopedic and urologic surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Ultrasound View | 10 minutes
  Ultrasound visibility of Dura Mater complexes on the intervertebral space chosen for spinal anesthesia
Difficulty in performing spinal anesthesia | 20 minutes
  Difficult spinal anesthesia includes: failure, procedure lasting more than 400 seconds from the insertion of the needle to the deliquoration; a number of needle replacements greater than 10; a change of the clinician practicing spinal anesthesia.

SECONDARY OUTCOMES:
Failure Rate | 20 minutes
  Failed Spinal Anesthesia
Duration | 20 minutes
  Spinal anesthesia duration (expressed in seconds) from the insertion of the needle to the deliquoration
Spinal needle replacements | 20 minutes
  Number of needle replacements

CONTACTS AND LOCATIONS:
Overall Officials: Felice E Agrò, Prof., Study Chair — Campus Biomedico of Rome
Locations (1):
- Università Campus Biomedico, Roma, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chin KJ, Ramlogan R, Arzola C, Singh M, Chan V. The utility of ultrasound imaging in predicting ease of performance of spinal anesthesia in an orthopedic patient population. Reg Anesth Pain Med. 2013 Jan-Feb;38(1):34-8. doi: 10.1097/AAP.0b013e3182734927. PMID 23143015
- [Background] Weed JT, Taenzer AH, Finkel KJ, Sites BD. Evaluation of pre-procedure ultrasound examination as a screening tool for difficult spinal anaesthesia*. Anaesthesia. 2011 Oct;66(10):925-30. doi: 10.1111/j.1365-2044.2011.06834.x. Epub 2011 Jul 25. PMID 21790522
- [Background] Del Buono R, Pascarella G, Costa F, Terranova G, Leoni ML, Barbara E, Carassiti M, Agro FE. Predicting difficult spinal anesthesia: development of a neuraxial block assessment score. Minerva Anestesiol. 2021 Jun;87(6):648-654. doi: 10.23736/S0375-9393.20.14892-2. Epub 2020 Dec 16. PMID 33325214